CLINICAL TRIAL: NCT02199223
Title: Combination Study of Panitumumab and Regorafenib in Advanced or Metastatic KRAS and NRAS Wild Type Colorectal Cancers
Brief Title: Regorafenib + Panitumumab for Colorectal Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI72561
Record Dates: First submitted 2014-06-30; First posted 2014-07-24 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: KRAS and NRAS Wild-type Colorectal Cancer
MeSH Terms: interventions — regorafenib; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- panitumumab + regorafenib (Experimental)
  Interventions: Drug: regorafenib + panitumumab

INTERVENTIONS:
Drug: regorafenib + panitumumab

SUMMARY:
Evaluate the safety of regorafenib and panitumumab

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of un-resectable or metastatic colorectal cancer which is KRAS and NRAS mutation negative (wild-type). Patients with any known mutation in KRAS or NRAS codons 12, 13, 59, 61, 117 or 146 will be excluded. Mutations of KRAS and NRAS codons not listed above are allowed. Biopsy of metastatic lesion is not required.
* Patients must show signs of progression (by imaging, or tumor marker elevation) after being treated with a first line or greater treatment for their un-resectable or metastatic colorectal cancer.
* Age 18 years or older.
* ECOG Performance Status 0-1
* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* Acute toxic effects of all prior treatment have resolved to NCI-CTCAE v4.0 less than or equal to Grade 1 or baseline prior to beginning treatment. Alopecia (any grade) is allowed. Peripheral neuropathy less than or equal to Grade 2 is allowed.
* Adequate bone marrow, renal and liver function as assessed by protocol laboratory requirements
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the ICF until at least 3 months after the last dose of study drug. Highly effective contraception must be used (e.g. male condom with spermicidal, diaphragm with spermicidal, intra-uterine device) must be used by both sexes.
* Subject must be able to swallow medication.
* Measurable disease at screening by RECIST 1.1 criteria

Exclusion Criteria:

* Any known mutation in KRAS or NRAS codons 12, 13, 59, 61, 117 or 146.
* Prior use of regorafenib.
* Known or suspected grade 3 allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of the trial.
* Uncontrolled hypertension (systolic pressure greater than140 mm Hg or diastolic pressure greater than 90 mm Hg [NCI-CTCAE v4.0] on mean of 3 consecutive readings despite optimal medical management. Hypertension may be corrected by adding or adjusting anti-hypertensives prior to the initiation of treatment at the discretion of the practitioner.
* Active or clinically significant cardiac disease including congestive heart failure, uncontrolled cardiac arrhythmias, or unstable angina.
* Evidence or history of congenital or acquired hypocoagulability disorders.
* Any hemorrhage or bleeding event greater than or equal to NCI CTCAE v.4.0 Grade 3 within 4 weeks prior to start of study medication.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism that have initiated within 6 months of start of study treatment. Stable, persistent events under appropriate management diagnosed greater than 6 months prior to treatment are allowed at the discretion of the investigator.
* Subjects who are receiving treatment for a concurrent cancer that is distinct in primary site or histology from colorectal carcinoma, except any cancer in-situ, treated basal cell or squamous cell carcinoma, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease more than 1 year before randomization are allowed. All cancer treatments must be completed at least 1 year prior to start of study treatment.
* Patients with severe hepatic impairment (Child-Pugh Class C).
* Known history of human immunodeficiency virus (HIV) infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy. Baseline testing is not required.
* Patients requiring IV antiviral or IV antibiotic treatment for ongoing infections.
* Symptomatic metastatic brain or meningeal tumors. Baseline brain imaging is not required.
* Presence of a non-healing wound or bone fracture.
* Patient's with a history of kidney disease or persistent proteinuria must have less than Grade 3 proteinuria per NCI CTCAE v4.0 at screening. If a patient has a history of kidney disease or persistent proteinuria, a urine protein test will be performed on a random urine sample. If the result is normal then no additional testing is required. If the result is abnormal, a 24 hour urine will be collected to determine if proteinuria is less than Grade 3.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Any malabsorption condition that in the opinion of the investigator would significantly impact drug absorption.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that in the opinion of the investigator may interfere with the subject's participation in the study or evaluation of the study results.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) within 3 weeks of starting study treatment.
* Concurrent use of another investigational drug or device during, or within 3 weeks of starting study treatment.
* Major surgical procedure, open biopsy, or significant traumatic injury within 3 weeks before start of study medication.
* Concurrent use of strong CYP3a4 inducers (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort)
* Concurrent use with strong inhibitors of CYP3A4 (e.g. clarithromycin, grapefruit juice, itraconazole, ketoconazole, nefazadone, posaconazole, telithromycin, and voriconazole)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety of regorafenib + panitumumab | Safety of the drug combination will be measured by number and severity of adverse events experienced while patients are on treatment which will be about 2-3 months if not more depending on the response to treatment.
  safety of combination for duration of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States